CLINICAL TRIAL: NCT01154322
Title: Pediatric Nasal Mask Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-09-09
Record Dates: First submitted 2010-06-15; First posted 2010-06-30 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pediatric mask (Experimental)
  Interventions: Device: Pixi pediatric mask

INTERVENTIONS:
Device: Pixi pediatric mask — The study mask is designed for use with PAP therapy to treat OSA in pediatric patients aged 2-7 years. The study mask is designed to be used in the hospital and the home environment. The study subject will use the device for up to 30 days while participating in the study.

SUMMARY:
The purpose of the study is to demonstrate the effectiveness of a pediatric mask in treating obstructive sleep apnea (OSA) in a pediatric population.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a condition in which there is partial or complete collapse of the upper airway during sleep. Features of OSA include snoring to upper airway resistance, which could be mild to severe. While OSA has been studied extensively in an adult population, research indicates that OSA is prevalent in a pediatric population as well, though the options for treatment are not as varied as that for the adult population. The study seeks to determine if a mask made for a pediatric population effectively treats their OSA.

ELIGIBILITY:
Inclusion Criteria:

* 2-7 years of age
* Diagnosis of OSA
* Current PAP therapy user
* Current nasal mask user

Exclusion Criteria:

* Recent sinus surgery
* Allergies to mask material
* Current seasonal allergies that could interfere with therapy
* History of clinically significant epistaxis in past 6 months
* Upper airway surgery less than 60 days before study entry

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford Center for Human Sleep Research, Redwood City, California
  - The Children's Hopsital, Aurora, Colorado
  - Gaylord Sleep Medicine, Wallingford, Connecticut

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric Mask: Pixi pediatric mask : The study mask is designed for use with PAP therapy to treat OSA in pediatric patients aged 2-7 years. The study mask is designed to be used in the hospital and the home environment. The study subject will use the device for up to 30 days while participating in the study.
Period: Overall Study
Arm/Group | Pediatric Mask
Started | 16
Completed | 14
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pediatric Mask
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index (AHI) Using the New Pediatric Mask (Pixi) Compared to the Child's Currently-used Mask
Description: Apnea-Hypopnea index (AHI) is an average of the number of apneas and hypopneas that occur over an hour of recorded sleep. AHI quantifies the severity of sleep disordered breathing (SDB). The higher the AHI, the more severe the SDB (mild 5-15, moderate 15-30, severe >30). In clinical practice an AHI <5 demonstrates efficacy of treatment. AHI was recorded during a monitored sleep study on the new Pixi mask, and compared with the AHI from a monitored sleep study on the child's usual mask. The outcome hypothesis was that the Pixi mask AHI would be equivalent or reduced compared to the child's usual mask.
Time Frame: Baseline AHI
Population: Subjects who completed all visits and procedures
Measure: Mean (Standard Deviation); unit: AHI (events/hour)
Groups:
- Currently-used Mask: Baseline AHI prior to Pixi mask use
Arm/Group | Currently-used Mask
Number analyzed (Participants) | 14
AHI (events/hour) | 2.7 (5.6)

2. Primary Outcome: Apnea-Hypopnea Index (AHI) Using the New Pediatric Mask (Pixi) Compared to the Child's Currently-used Mask
Description: Apnea-Hypopnea index (AHI) is an average of the number of apneas and hypopneas that occur over an hour of recorded sleep. AHI quantifies the severity of sleep disordered breathing (SDB). The higher the AHI, the more severe the SDB (mild 5-15, moderate 15-30, severe >30). In clinical practice an AHI <5 demonstrates efficacy of treatment. AHI was recorded during a monitored sleep study on the new Pixi mask and compared with the AHI from a monitored sleep study on the child's usual mask. The outcome hypothesis was that the Pixi mask AHI would be equivalent or reduced compared to the child's usual mask.
Time Frame: AHI after min 21 days use with Pixi mask
Measure: Mean (Standard Deviation); unit: AHI (events/hour)
Groups:
- Pixi Mask: AHI with Pixi mask
Arm/Group | Pixi Mask
Number analyzed (Participants) | 14
AHI (events/hour) | 1.2 (1.5)

ADVERSE EVENTS:
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=16)
Seizure (Nervous system disorders) | 1 (1) — Seizure unrelated to use of PAP/Pixi mask

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less